CLINICAL TRIAL: NCT06053710
Title: Detecting Local and Systemic Fluid Accumulation With a Wearable Bioimpedance Sensor in Patients With Fluid Management Problems (DELOS)
Brief Title: Detecting Fluid Accumulation With a Wearable Bioimpedance Sensor
Acronym: DELOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mode Sensors AS (Industry)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTR0042A DELOS
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Overhydration; Kidney Failure; Edema
Keywords: Hydration
MeSH Terms: conditions — Water Intoxication; Renal Insufficiency; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with chronic kidney failure (Other): Patients with chronic kidney failure will wear bioimpedance sensors at the upper back and lower anterior leg for three weeks.
  Interventions: Device: Wearable bioimpedance sensor
- Patients with severe overhydration (Other): Patients with severe overhydration will wear bioimpedance sensors at the upper back, lateral thorax, anterior thigh, and lower anterior leg throughout an intensive dialysis treatment regime (~2-10 days).
  Interventions: Device: Wearable bioimpedance sensor

INTERVENTIONS:
Device: Wearable bioimpedance sensor — The investigational device is an electronic bioimpedance-based, body-worn, battery-powered sensor intended to monitor changes in fluid volume. It is designed as an adhesive patch with four integrated electrodes.

SUMMARY:
The investigation is a prospective cohort study, where two patient groups will be monitored by a wearable bioimpedance sensor during their scheduled treatment. The overall objective is to assess the bioimpedance sensor's ability to detect local and systemic fluid accumulation.

Sub-investigation A will investigate the ability of the device to detect fluid accumulation in patients with stable chronic kidney disease undergoing regular and planned hemodialysis.

Sub-investigation B will investigate the ability of the device to track hydration status in patients scheduled for an "intensive" dialysis treatment regime, due to severe overhydration.

DETAILED DESCRIPTION:
In Sub-investigation A, patients will be monitored for at least 10 consecutive dialysis sessions, and for a minimum of 3 weeks. Patients will wear two sensors (upper back and lower anterior leg).

In Sub-investigation B, patients will use the device throughout their whole treatment period, and for most patients, this will correspond to 2-6 dialysis treatments over 3 to 10 days. Patients will wear four patches (upper back, lateral thorax, anterior thigh, and lower anterior leg).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Regular hemodialysis (≥ 2 times weekly) with ultrafiltration volume ≥ 1 liter (Sub-investigation A)
* Scheduled for intensive dialysis treatment due to severe overhydration (Sub-investigation B)

Exclusion Criteria:

* Known allergies or skin sensitivities to electrode hydrogel and/or acrylic adhesives
* Implantable pulse generators such as pacemakers and defibrillators, and/or use of other electrical medical equipment for which an interaction effect with the investigational device cannot be ruled out.
* Patients undergoing MRI
* Breached skin at patch mounting area
* Pregnancy
* Any medical or psychiatric condition, which in the opinion of the investigator precludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of interdialytic fluid accumulation on the extracellular resistance of the upper back in stable chronic dialysis patients | 1-4 days
  Relative change in extracellular resistance of the upper back, measured by the bioimpedance device in the interdialytic period in Sub-investigation A

SECONDARY OUTCOMES:
The effect of interdialytic fluid accumulation on the extracellular resistance of the lower anterior leg in stable chronic dialysis patients | 1-4 days
  Relative change in extracellular resistance of the lower anterior leg, measured by the bioimpedance device in the interdialytic period in Sub-investigation A
The effect of an intensive dialysis treatment regime on the extracellular resistance of the upper back in patients with severe overhydration | 2-10 days
  Relative change in extracellular resistance of the upper back, measured by the bioimpedance device from before to after the dialysis treatment regime in Sub-investigation B
The effect of an intensive dialysis treatment regime on the extracellular resistance of the lower anterior leg in patients with severe overhydration | 2-10 days
  Relative change in extracellular resistance of the lower anterior leg, measured by the bioimpedance device from before to after the dialysis treatment regime in Sub-investigation B
The effect of an intensive dialysis treatment regime on the extracellular resistance of the lateral thorax in patients with severe overhydration | 2-10 days
  Relative change in extracellular resistance of the lateral thorax, measured by the bioimpedance device from before to after the dialysis treatment regime in Sub-investigation B
Safety of the investigational device | Up to 4 weeks
  Frequency and severity of adverse device effects.
The effect of an intensive dialysis treatment regime on the extracellular resistance of the anterior thigh | 2-10 days
  Relative change in extracellular resistance of the anterior thigh, measured by the bioimpedance device

CONTACTS AND LOCATIONS:
Overall Officials: Sigve N Aas, PhD, Study Director — Mode Sensors AS; Nanna von der Lippe, PhD, Principal Investigator — Oslo University Hospital; Hege K Pihlstrøm, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Rikshospitalet, Oslo University Hospital, Oslo
  - Ullevål sykehus, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No